CLINICAL TRIAL: NCT03250936
Title: Descriptive Study of Trampoline Accidents in the Pediatric Emergency Department of Rennes
Acronym: TRAUMPO
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC16_3058
Record Dates: First submitted 2017-08-11; First posted 2017-08-16 (Actual); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Trauma; Emergencies; Child, Only
Keywords: trampoline
MeSH Terms: conditions — Wounds and Injuries; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Trampoline group: Child patients with trauma due to trampoline from june 2016 to december 2016 consulting in emergencies unit of Rennes' hospital
- Control group: Child patients with trauma related to sport from june 2016 to december 2016 consulting in emergencies unit of Rennes' hospital

SUMMARY:
The aim of this study is to compare trauma related to others sport to trauma due to trampoline in pediatric emergencies of Rennes.

DETAILED DESCRIPTION:
Trampoline accidents are increasing since a few years. In Rennes hospital, pediatric emergencies are experiencing a subjective increase in admissions for trampoline trauma with increasingly early ages and severe trauma. The aim of this study is to compare trauma related to others sport to trauma due to trampoline in pediatric emergencies of Rennes.

In parallel, retrospective data analysis will be performed on the same data during the year 2008, to compare with a period before the explosion of trampoline sales.

ELIGIBILITY:
Inclusion Criteria:

* Child from 2 to 16 years old
* Childs admitted in emergencies unit for a trauma
* Parents not opposed in their child's participation to the study

Exclusion Criteria:

* Child under 2 years old (before learning to walk)
* Single wounds and head injuries not related to sports activities (Fall from a bed or from its height, simple wound with sharp objects)

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children between 2 and 16 years old consulting in pediatric emergencies for a trauma related to trampoline Children between 2 and 16 years old consulting in pediatric emergencies for a trauma related to others sport
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2016-12-06 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Types of trauma related to trampoline compared to trauma related to others sport in pediatric emergencies of Rennes. | 6 months
  Types of trauma related to trampoline compared to trauma related to others sport in pediatric emergencies of Rennes.

SECONDARY OUTCOMES:
Arguments for preventive management in the general practitioner | 6 months
  Arguments for preventive management in the general practitioner

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Fraisse, Dr, Principal Investigator — Rennes University Hospital
Locations (1):
- Pediatric and orthopedic surgery division, Rennes, France